CLINICAL TRIAL: NCT02179892
Title: Comparison Between Bupivacaine Extended-Release Liposome Injection (Exparel) Versus Bupivacaine With Dexamethasone in Transversus Abdominis Plane Block: A Prospective Randomized Controlled Trial
Brief Title: Comparison of Exparel to Bupivacaine With Dexamethasone in TAP Block
Acronym: TapBlock
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate patient population to complete enrollment
Sponsor: Colette Curtis MD (Other)
Responsible Party: Sponsor-Investigator, Colette Curtis MD, Assistant Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00071635
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Pain
Keywords: anesthesia; surgery; pain
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Calcium Dobesilate; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1-Exparel (Active Comparator): Bupivacaine Extended-Release Liposome Injection (Exparel)will be administered via TAP block procedure
  Interventions: Drug: Bupivacaine Extended-Release Liposome Injection (Exparel); Drug: IV Acetaminophen; Drug: Oral Acetaminophen
- Group 2-Bupivacaine and Dexamethasone IV (Active Comparator): Bupivacaine and Dexamethasone Injection will be administered via TAP block procedure.
  Interventions: Drug: Bupivacaine and Dexamethasone Injection; Drug: IV Acetaminophen; Drug: Oral Acetaminophen

INTERVENTIONS:
Drug: Bupivacaine Extended-Release Liposome Injection (Exparel) — 266mg/30mL of Exparel will be injected via unilateral TAP block
  Arms: Group 1-Exparel
Drug: Bupivacaine and Dexamethasone Injection — As a combination injection, 28 ml of 0.375% bupivacaine and 8 mg/2ml of dexamethasone will be injected via unilateral TAP block.
  Arms: Group 2-Bupivacaine and Dexamethasone IV
Drug: IV Acetaminophen — Intravenous (IV) acetaminophen 1000 mg every 8 hours for 8 doses.
Drug: Oral Acetaminophen — Oral acetaminophen 650 mg every 6 hours.

SUMMARY:
The purpose of this study is to compare the efficacy and duration of bupivacaine extended-release liposome injection (Exparel) versus bupivacaine with dexamethasone in transversus abdominis plane (TAP) blocks for patients undergoing abdominal surgery at Emory University Hospital and Emory University Hospital Midtown.

The investigators hypothesize that Exparel will provide greater postoperative pain relief than bupivacaine with dexamethasone. The investigators plan to enroll up to 50 male and female subjects meeting inclusion and exclusion criteria who will be randomized to receive either Exparel (Group 1) or bupivacaine with epinephrine and dexamethasone (Group 2) in the TAP block to achieve at least 22 subjects in each group

DETAILED DESCRIPTION:
Group 1 will be administered 266 mg of Exparel, diluted to 30 mL. Group 2 will be given 28 mL of 0.375% bupivacaine and 8mg/2 mL dexamethasone.Before injection of the study medication, 2mL of normal saline with be injected under ultrasound visualization to ensure needle tip is in the transversus abdominis plane.Randomization will occur following the written informed consent and prior to the start of the surgical procedure. Postoperatively, study patients will receive intravenous acetaminophen 1000mg every 8 hours for 3 doses, then oral acetaminophen 650mg every 6 hours. Subjects will also have patient-controlled analgesia (PCA) with morphine or hydromorphone. The research staff recording data will be blinded to the treatment group. Demographic data will be recorded, including age, date of birth, height and weight to ensure similarity between the two groups. A medical history will be obtained as well as surgical and anesthesia details. Study patients will be followed for 72 hours postoperatively to record the amount of opioid consumption, as well as other pain score data using the Visual Analogue Scale (VAS).The subject's participation will end 72 hours after surgery. A telephone interview will occur with the subject if hospital discharge occurs prior to 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients undergoing scheduled abdominal surgery at Emory University Hospital or Emory University Hospital Midtown
* Patients willing and able to provide written informed consent

Exclusion Criteria:

* Patients less than 18 years of age, since Exparel has not been studied in this age group
* Patients who are pregnant or lactating, since Exparel has not been shown to be safe in this population, and because of potential drug transfer to child
* Patients with uncontrolled diabetes since dexamethasone may cause hyperglycemia
* Patients with liver dysfunction, since bupivacaine is hepatically metabolized
* Patients with renal failure, since bupivacaine is renally excreted, defined as requiring hemodialysis or renal replacement therapy
* Patients with allergy to one of the study drugs
* Patients with local infection, which may be exacerbated by dexamethasone
* Patients with significant opioid tolerance, defined as taking at least 60 mg oral morphine per day, 3 mg oral oxycodone per day, 25 mcg/hr fentanyl patch, 25 mg oral oxymorphone per day, 8 mg of oral hydromorphone per day or an equianalgesic dose of another opioid for one week or longer
* Patients with known coagulopathy, since bleeding risk is higher Patients who are getting neuraxial anesthesia for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06-06 (Actual); Study Completion 2015-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette Curtis, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory University Hospital and the Emory University Hospital Midtown between July 2014 through June 2015.
Groups:
- Group 1-Exparel: Bupivacaine Extended-Release Liposome Injection (Exparel) were administered via TAP block procedure
  Bupivacaine Extended-Release Liposome Injection (Exparel): 266mg/30mL of Exparel was injected via unilateral TAP block.
- Group 2-Bupivacaine and Dexamethasone IV: Bupivacaine and Dexamethasone Injection were administered via TAP block procedure.
  Bupivacaine and Dexamethasone Injection: As a combination injection, 28 ml of 0.375% bupivacaine and 8 mg/2ml of dexamethasone was injected via unilateral TAP block.
Period: Overall Study
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1-Exparel: Bupivacaine Extended-Release Liposome Injection (Exparel) was administered via TAP block procedure
  Bupivacaine Extended-Release Liposome Injection (Exparel): 266mg/30mL of Exparel was injected via unilateral TAP block
- Group 2-Bupivacaine and Dexamethasone IV: Bupivacaine and Dexamethasone Injection was administered via TAP block procedure.
  Bupivacaine and Dexamethasone Injection: As a combination injection, 28 ml of 0.375% bupivacaine and 8 mg/2ml of dexamethasone was injected via unilateral TAP block.
- Total: Total of all reporting groups
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Opioid Consumption
Description: The investigators will collect the total amount of opioid consumption for the 72 hour post operative period in each group.
Time Frame: Post Surgery (Up to 72 Hours)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV
Number analyzed (Participants) | 5 | 4
milligrams | 507 (602) | 392 (133)

2. Secondary Outcome: Mean Visual Analogue Scale (VAS) Pain Score at Rest
Description: The VAS method of pain assessment (scale of 1- 10) will be used to measure the participant's pain level at rest each day during the 72 hours post surgical period. One represents the lowest level of pain and 10 represents the highest level of pain.
Time Frame: Post-Surgery 24 Hours, 48 Hours, 72 Hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV
Number analyzed (Participants) | 5 | 4
units on a scale
  24 Hours Post Surgery | 4.2 (1.9) | 3.5 (1.3)
  48 Hours Post Surgery | 1.8 (1.6) | 3.3 (2.6)
  72 Hours Post Surgery | 1.8 (2.0) | 3.5 (2.6)

3. Secondary Outcome: Mean Visual Analogue Scale (VAS) Pain Score With Movement
Description: The VAS method of pain assessment (scale of 1-10) will be used to measure the patient's level of pain with movement each day during the 72 hour post surgical period. One represents the lowest level of pain and 10 represents the highest level of pain.
Time Frame: Post-Surgery 24 Hours, 48 Hours, 72 Hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV
Number analyzed (Participants) | 5 | 4
units on a scale
  24 Hours Post Surgery | 6.8 (3.4) | 5.8 (1.7)
  48 Hours Post Surgery | 6.6 (4.1) | 6.3 (3.3)
  72 Hours Post Surgery | 3.6 (2.9) | 4.8 (2.9)

4. Secondary Outcome: Mean Time of First Opioid Use
Description: The time of first opioid use after surgery will be recorded for up to 72 hours.
Time Frame: Post-surgery (Up to 72 Hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV
Number analyzed (Participants) | 5 | 4
hours | 58 (29) | 46 (31)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (1 year).
Arm/Group | Group 1-Exparel | Group 2-Bupivacaine and Dexamethasone IV
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes